CLINICAL TRIAL: NCT01467037
Title: Vaccine Effectiveness of RV1 in a Naïve Population
Status: Completed | Type: Observational
Sponsor: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Collaborators: Institut National en Santé Publique du Québec (Other); Ministere de la Sante et des Services Sociaux (Other); GlaxoSmithKline (Industry)
Responsible Party: Principal Investigator, Caroline Quach-Thanh, MD, MSc, FRCPC, McGill University Health Centre/Research Institute of the McGill University Health Centre
Other Study IDs: MCH-ID-11-01
Record Dates: First submitted 2011-11-04; First posted 2011-11-08 (Estimated); Results first posted 2016-01-29 (Estimated); Last update posted 2016-04-19 (Estimated); Status verified 2016-03

CONDITIONS: Rotavirus Infections; Gastroenteritis; Diarrhea
Keywords: Rotavirus; Gastroenteritis; Vaccination; Pediatrics
MeSH Terms: conditions — Rotavirus Infections; Gastroenteritis; Diarrhea

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — stool sample
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Rotavirus-negative: Patients with a negative result for rotavirus via enzyme immunoassay (EIA). No intervention done.
  Interventions: Other: No intervention done
- Rotavirus-positive: Patients with a positive result for rotavirus via enzyme immunoassay (EIA). Rotavirus-positives were confirmed via real-time reverse-transcriptase polymerase chain reactions (RT-PCR). RT-PCR results were used in the event of discordant EIA results. Rotavirus genotyping was performed. No intervention done.
  Interventions: Other: No intervention done

INTERVENTIONS:
Other: No intervention done — Not applicable because no intervention was done.

SUMMARY:
Rotavirus (RV) is the leading cause of severe gastroenteritis (GE) in young children. The cumulative risk of GE hospitalizations and hospital stays of < 24 hours is 1/25, which would amount to 13,600 Canadian children < 5 years. The incidence of nosocomial RV infections is an average of 8/10,000 patient-days in children < 5 years. An immunization program with a live-attenuated monovalent oral RV vaccine (RV1 - Rotarix® from GSK) will be implemented, free of charge, in the Province of Quebec in November 2011. To provide an accurate portrait of the disease and give critical information to the public health agencies as they struggle to control costs, we aim to evaluate the accuracy of surveillance for RV and other diseases with similar characteristics; estimate selection bias in passive laboratory-based surveillance; and estimate the agreement between surveillance time-series created from passive and active surveillance data sources.

DETAILED DESCRIPTION:
In November 2011, Quebec implemented a publicly-funded RV1 vaccination program with its routine administration at 2 and 4 months of age. From February 1, 2012 - May 31, 2014, we conducted prospective, active surveillance for acute rotavirus gastroenteritis at The Montreal Children's Hospital and Centre Hospitalier Universitaire Sainte-Justine, located in Montreal, and Centre Hospitalier Universitaire de Sherbrooke, located in Sherbrooke. Active surveillance was approved by Research Ethics Boards at each hospital.

ELIGIBILITY:
Inclusion Criteria:

* Child less than 3 years old

Cases:

* Acute gastroenteritis (within 7 days of hospital visit)
* able to provide a stool specimen for RV ELISA testing
* Rotavirus positive

Controls:

* Visited the ED or admitted for a non-rotavirus gastroenteritis
* Visited the ED or admitted for acute respiratory infections without gastroenteritis symptoms

Exclusion Criteria:

* Immunocompromised children
* Prior history of intussusception
* Admission to NICU between 6 to 15 weeks of life, for >6 weeks
* Child less than 56 days of life (8 weeks)
* Child vaccinated with Rotateq (Merck)

Ages: 8 Weeks to 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: The Montreal Children's Hospital and the CHU Sainte-Justine are the 2 main pediatric hospitals in Montreal. With these 3 sites, 30% of the Quebec birth cohort will be captured and, given the concentration of children in the Montreal area, the participating hospitals will ensure that the study remains efficient in terms of resources. We elected Sherbrooke as an intermediate area; Montreal will represent an urban population.
Sampling Method: Non-Probability Sample
Enrollment: 374 (Actual)
Dates: Start 2012-02; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Caroline Quach-Thanh, MD, MSc, Principal Investigator — McGill University Health Centre/Research Institute of the McGill University Health Centre; Caroline Quach-Thanh, MD, MSc, Study Director — McGill University Health Centre/Research Institute of the McGill University Health Centre
Locations (3):
- Canada (3):
  - The Montreal Children's Hospital, Montreal, Quebec
  - Centre Hospitalier Universitaire Sainte-Justine, Montreal, Quebec
  - Centre Hospitalier Universitaire de Sherbrooke, Sherbrooke, Quebec

REFERENCES:
- [Result] Doll MK, Buckeridge DL, Morrison KT, Gagneur A, Tapiero B, Charest H, Quach C. Effectiveness of monovalent rotavirus vaccine in a high-income, predominant-use setting. Vaccine. 2015 Dec 16;33(51):7307-7314. doi: 10.1016/j.vaccine.2015.10.118. Epub 2015 Nov 3. PMID 26546262

RESULTS

PARTICIPANT FLOW:
Recruitment Details: We conducted prospective, active surveillance for acute rotavirus gastroenteritis at The Montreal Children's Hospital and Centre Hospitalier Universitaire Sainte-Justine, located in Montreal, and Centre Hospitalier Universitaire de Sherbrooke, located in Sherbrooke.
Groups:
- Vaccine Effectiveness Study Population: Among patients eligible for active surveillance of acute gastroenteritis, patients aged <15 months at RV1 program implementation (November 1, 2011), AND aged ≥16 weeks at symptom onset
Period: Overall Study
Arm/Group | Vaccine Effectiveness Study Population
Started | 374
Completed | 374
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Among all active surveillance eligible patients, patients were included if parent/legal guardian had provided informed consent, and if an adequate stool specimen was provided within 7 days of hospital presentation. Patients needed to be aged <15 months at RV1 program implementation (November 1, 2011), AND aged ≥16 weeks at symptom onset.
Groups:
- Rotavirus-negative: All stool samples were initially tested for rotavirus via enzyme immunoassay. Patients with a negative result are included in this group.
- Rotavirus -Positive: All stool were initially tested for rotavirus via enzyme immunoassay. Rotavirus-positives were confirmed via real-time reverse-transcriptase polymerase chain reactions (RT-PCR). RT-PCR results were used in the event of discordant EIA results. Rotavirus genotyping was performed.
- Total: Total of all reporting groups
Arm/Group | Rotavirus-negative | Rotavirus -Positive | Total
Number analyzed (Participants) | 342 | 32 | 374
Age, Continuous [Mean (Standard Deviation); unit: months] | 12.6 (6.3) | 16.6 (6.5) | 13 (6.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 154 | 20 | 174
  Male | 188 | 12 | 200
Region of Enrollment [Number; unit: participants]
  Canada | 342 | 32 | 374
Rotavirus vaccination [Number; unit: participants]
  RV-vaccination 0 dose | 62 | 24 | 86
  RV-vaccination 1-dose | 26 | 1 | 27
  RV-vaccination ≥2 doses | 254 | 7 | 261

OUTCOME MEASURES:

1. Primary Outcome: Matched VE Participants
Description: RV1 vaccine effectiveness (VE) was investigated using a subset of active surveillance participants age-eligible to receive 2-doses of RV1 vaccine, defined as participants (i) <15 weeks of age as of program implementation (November 1, 2011), and (ii) ≥16 weeks of age at symptom onset. These ages corresponded to the maximum recommended age of administration for the first RV1 dose at program implementation, and the recommended age of second dose administration, respectively.
  We estimated RV1 VE of 2- versus 0-doses and ≥1- versus 0-doseto prevent rotavirus hospitalization or emergency visits. Only valid RV1 vaccinations administered ≥14 days prior to symptom onset were considered. Children vaccinated with RV5 (private market,minimal penetrance) were excluded.
Time Frame: From February 1, 2012 to May 31, 2014
Population: Rotavirus vaccination history by rotavirus disease status among matched VE participants
Measure: Number; unit: participants
Groups:
- Rotavirus-positive: All stool were initially tested for rotavirus via enzyme immunoassay. Rotavirus positives were confirmed via realtime reversetranscriptase polymerase chain reactions (RTPCR). RTPCR results were used in the event of discordant EIA results. Rotavirus genotyping was performed.
Arm/Group | Rotavirus-negative | Rotavirus-positive
Number analyzed (Participants) | 156 | 30
participants
  0-Doses | 26 | 22
  1 Dose | 16 | 1
  2 Doses | 114 | 7

2. Other Pre Specified Outcome: Vaccine Effectiveness of RV1
Description: RV1 vaccine effectiveness (VE) was investigated using a subset of active surveillance participants age-eligible to receive 2-doses of RV1 vaccine, defined as participants (i) <15 weeks of age as of program implementation (November 1, 2011), and (ii) ≥16 weeks of age at symptom onset. These ages corresponded to the maximum recommended age of administration for the first RV1 dose at program implementation, and the recommended age of second dose administration, respectively.
  Only valid RV1 vaccinations administered ≥14 days prior to symptom onset were considered. RV1 VE was estimated as (1 - exposure odds ratio) × 100. Based upon our sampling scheme, the exposure odds ratio from our analyses approximates the rate ratio.
Time Frame: From February 1, 2012 to May 31, 2014
Measure: Number (95% Confidence Interval); unit: adjusted VE
Groups:
- 2 Versus 0 Doses: We compared Rotavirus VE between patients that received 2 versus 0 doses of RV1.
- ≥1 Versus 0 Dose: We compared Rotavirus VE between patients that received 1 versus 0 dose of RV1.
Arm/Group | 2 Versus 0 Doses | ≥1 Versus 0 Dose
Number analyzed (Participants) | 169 | 186
adjusted VE | 91.2 [61.6 to 98.0] | 92.5 [69.3 to 98.2]
Statistical Analysis 1: Comparison: 2 Versus 0 Doses; Test type: Superiority or Other; Adjusted OR = 0.088, 95% CI 2-sided [0.020 to 0.384] — Conditional logistic regression was used. Adjusted VE = (1 - adjusted OR) *100
Statistical Analysis 2: Comparison: ≥1 Versus 0 Dose; Test type: Superiority or Other; Adjusted OR = 0.075, 95% CI 2-sided [0.018 to 0.307] — Conditional logistic regression was used. Adjusted VE = (1 - adjusted OR) *100

ADVERSE EVENTS:
Description: Adverse events were not collected. We did not administer any medication nor vaccine.
Arm/Group | Vaccine Effectiveness Study Population
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No